CLINICAL TRIAL: NCT04674813
Title: A Phase 1, Multicenter, Open-Label Study of CC-95266 in Subjects With Relapsed and/or Refractory Multiple Myeloma
Brief Title: A Study of CC-95266 in Participants With Relapsed and/or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Juno Therapeutics, a Subsidiary of Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-95266-MM-001; U1111-1260-4921 (Registry Identifier: WHO)
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma
Keywords: CC-95266; Multiple Myeloma; Relapsed and/or Refractory
MeSH Terms: conditions — Multiple Myeloma | interventions — fludarabine; Cyclophosphamide; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Administration of CC-95266 (Experimental)
  Interventions: Drug: CC-95266; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Bendamustine

INTERVENTIONS:
Drug: CC-95266 — Specified dose on specified days
Drug: Fludarabine — Specified dose on specified days
Drug: Cyclophosphamide — Specified dose on specified days
Drug: Bendamustine — Specified dose on specified days

SUMMARY:
The purpose of this study is to evaluate the safety and preliminary efficacy of CC-95266 in participants with relapsed and/or refractory multiple myeloma (R/R MM).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Participant has a diagnosis of multiple myeloma (MM) with relapsed and/or refractory disease. Participants must have confirmed progressive disease (as per IMWG criteria) on or within 12 months of completing treatment with the last anti-myeloma treatment regimen before study entry or have confirmed progressive disease within 6 months prior to screening and who are subsequently determined to be refractory or non-responsive to their most recent anti-myeloma treatment regimen, except for participants with cellular therapy (e.g., Chimeric antigen receptor (CAR) T-cell therapy) as their last treatment, who may enroll beyond 12 months.
* Participants in Part A, and Part B Cohort A, and Part B Cohort B must have received at least 3 prior anti-myeloma treatment regimens (note: induction with or without hematopoietic stem cell transplant (HSCT) and with or without maintenance therapy is considered one regimen).Subjects in Part B Cohort C only must have received at least 1 but not greater than 3 prior anti-myeloma treatment regimens, including a proteasome inhibitor and immunomodulatory agent including:

  * Autologous HSCT, unless the subject was ineligible
  * A regimen that included an immunomodulatory agent (e.g., thalidomide, lenalidomide, pomalidomide) and a proteasome inhibitor (e.g., bortezomib, carfilzomib, ixazomib), either alone or combination
  * Anti-CD38 (e.g., daratumumab), either alone or combination. Subjects in Cohort C do not require prior anti-CD38 antibody therapy.
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ function

Exclusion Criteria:

* Known active or history of central nervous system (CNS) involvement of MM
* Active or history of plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, skin changes) syndrome, or clinically significant amyloidosis
* Active autoimmune disease requiring immunosuppressive therapy
* History or presence of clinically significant CNS pathology such as seizure disorder, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, or psychosis

Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2025-12-22 (Actual); Study Completion 2025-12-22 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Up to 2 years after CC-95266 infusion
Number of participants with significant laboratory abnormalities | Up to 2 years after CC-95266 infusion
Number of participants with Dose Limiting Toxicities (DLTs) | Up to 2 years after CC-95266 infusion
Maximum Tolerated Dose (MTD) | Up to 2 years after CC-95266 infusion
Recommended Phase 2 Dose (RP2D) | Up to 2 years after CC-95266 infusion

SECONDARY OUTCOMES:
Pharmacokinetics - Maximum plasma concentration of drug (Cmax) | Up to 2 years after CC-95266 infusion
Pharmacokinetics - Time to peak (maximum) serum concentration (tmax) | Up to 2 years after CC-95266 infusion
Pharmacokinetics - Area under the curve for days 1-29 after CC-95266 infusion (AUC1-29) | Up to 2 years after CC-95266 infusion
Overall response rate (ORR) | Up to 2 years after CC-95266 infusion
Complete response rate (CRR) | Up to 2 years after CC-95266 infusion
Very good partial response (VGPR) or better | Up to 2 years after CC-95266 infusion
Duration of response (DOR) | Up to 2 years after CC-95266 infusion
Duration of complete response (DOCR) | Up to 2 years after CC-95266 infusion
Time to response (TTR) | Up to 2 years after CC-95266 infusion
Time to complete response (TTCR) | Up to 2 years after CC-95266 infusion
Progression-free survival (PFS) | Up to 2 years after CC-95266 infusion
Overall survival (OS) | Up to 2 years after CC-95266 infusion

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (10):
- United States (10):
  - Local Institution - 005, Birmingham, Alabama
  - Local Institution - 009, Duarte, California
  - Local Institution - 012, San Francisco, California
  - Local Institution - 002, Denver, Colorado
  - Local Institution - 008, Baltimore, Maryland
  - Local Institution - 010, Boston, Massachusetts
  - Local Institution - 011, New York, New York
  - Local Institution - 001, Nashville, Tennessee
  - Local Institution - 006, Dallas, Texas
  - Local Institution - 003, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com